CLINICAL TRIAL: NCT06335095
Title: Gait Analysis and Degenerative Spine
Status: Recruiting | Type: Observational
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Other Study IDs: a319
Record Dates: First submitted 2023-11-30; First posted 2024-03-28 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Spinal Disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy volunteers
  Interventions: Other: Kinematic sensors
- Disease
  Interventions: Other: Kinematic sensors

INTERVENTIONS:
Other: Kinematic sensors — Comparative analysis of kinematic data acquired in supervised and unsupervised environment

SUMMARY:
The goal of this observational study is to analyse the biomechanics of a degenerative spinal disease. The main questions it aims to answer are:

* What are the biomechanical variables affected by the disease
* How they evolve with disease progression and treatment

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 85 years
* Diagnosis of spinal disease by clinical and imagiological criteria
* More than 3 months duration of disease
* Ability to give consent
* Fluent portuguese speaker

Exclusion Criteria:

* Previous spine surgery
* Spinal instability
* Neurological disease that might interfere with walking
* Known orthopedic conditions that causes significant gait impairment
* Dementia or development disorder with cognitive impairment
* Inability to give consent

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of the spinal disease in study and that meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in gait parameter - speed (m/s) - at 3 months | 3 months
  The change will be defined by a 10% increase in speed (meters/second) at 3 months from baseline assessment.
Change from baseline in gait parameter - speed (m/s) - at 6 months | 6 months
  The change will be defined by a 10% increase in speed (meters/second) at 6 months from baseline assessment.
Change from baseline in gait parameter - speed (m/s) - at 12 months | 12 months
  The change will be defined by a 10% increase in speed (meters/second) at 12 months from baseline assessment.
Change from baseline in gait parameter - step length (m) - at 3 months | 3 months
  The change will be defined by a 10% increase in step length (meters) at 3 months from baseline assessment.
Change from baseline in gait parameter - step length (m) - at 6 months | 6 months
  The change will be defined by a 10% increase in step length (meters) at 6 months from baseline assessment.
Change from baseline in gait parameter - step length (m) - at 12 months | 12 months
  The change will be defined by a 10% increase in step length (meters) at 12 months from baseline assessment.
Change from baseline in gait parameter - step width (m) - at 3 months | 3 months
  The change will be defined by a 10% decrease in step width (meters) at 3 months from baseline assessment.
Change from baseline in gait parameter - step width (m) - at 6 months | 6 months
  The change will be defined by a 10% decrease in step width (meters) at 6 months from baseline assessment.
Change from baseline in gait parameter - step width (m) - at 12 months | 12 months
  The change will be defined by a 10% decrease in step width (meters) at 12 months from baseline assessment.

SECONDARY OUTCOMES:
Change from baseline in Back Pain as measured by the Numeric Pain Rating Scale (NPRS) at 3 months | 3 months
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥2 point in NRPS (range: 0 - 10 points).
Change from baseline in Back Pain as measured by the Numeric Pain Rating Scale (NPRS) at 6 months | 6 months
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥2 point in NRPS (range: 0 - 10 points).
Change from baseline in Back Pain as measured by the Numeric Pain Rating Scale (NPRS) at 12 months | 12 months
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥2 point in NRPS (range: 0 - 10 points).
Change from baseline in disability as measured by the Oswestry Disability Index (ODI) at 3 months | 3 months
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥27% in ODI (range: 0-50 and higher scores are indicative of more disability).
Change from baseline in disability as measured by the Oswestry Disability Index (ODI) at 6 months | 6 months
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥27% in ODI (range: 0-50 and higher scores are indicative of more disability).
Change from baseline in disability as measured by the Oswestry Disability Index (ODI) at 12 months | 12 months
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥27% in ODI (range: 0-50 and higher scores are indicative of more disability).
Change from baseline in Quality of Life as measured by the European Quality of Life-5 Dimensions Questionnaire (EQ-5D) at 3 months | 3 months
  Change from baseline in Quality of Life as measured by the European Quality of Life-5 Dimensions Questionnaire (EQ-5D) at 3 months
Change from baseline in Quality of Life as measured by the European Quality of Life-5 Dimensions Questionnaire (EQ-5D) at 6 months | 6 months
  Change from baseline in Quality of Life as measured by the European Quality of Life-5 Dimensions Questionnaire (EQ-5D) at 6 months
Change from baseline in Quality of Life as measured by the European Quality of Life-5 Dimensions Questionnaire (EQ-5D) at 12 months | 12 months
  Change from baseline in Quality of Life as measured by the European Quality of Life-5 Dimensions Questionnaire (EQ-5D) at 12 months
Change from baseline in disability as measured by the Core Outcome Measures Index (COMI) at 3 months | 3 months
  In the core COMI-back, 1 question consists of 2 numerical rating scales to be answered from 0 to 10 and 5 questions to be answered by selecting 1 of 5 response options. The average of the 2 disability scores forms the disability dimension subscore. A total COMI score is determined by averaging the 5 dimension scores.
Change from baseline in disability as measured by the Core Outcome Measures Index (COMI) at 6 months | 6 months
  In the core COMI-back, 1 question consists of 2 numerical rating scales to be answered from 0 to 10 and 5 questions to be answered by selecting 1 of 5 response options. The average of the 2 disability scores forms the disability dimension subscore. A total COMI score is determined by averaging the 5 dimension scores.
Change from baseline in disability as measured by the Core Outcome Measures Index (COMI) at 12 months | 12 months
  In the core COMI-back, 1 question consists of 2 numerical rating scales to be answered from 0 to 10 and 5 questions to be answered by selecting 1 of 5 response options. The average of the 2 disability scores forms the disability dimension subscore. A total COMI score is determined by averaging the 5 dimension scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital da Luz Setúbal, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided